CLINICAL TRIAL: NCT04416867
Title: A Comparison of the Efficacy of Physical Therapy and Radial Extracorporeal Shock Wave Therapy in the Treatment of Carpal Tunnel Syndrome: a Randomized Control Study
Brief Title: Radial Extracorporeal Shock Wave Therapy in the Treatment of Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Regional Training & Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gonca Saglam, Head of Physical medicine and rehabilitation department, Erzurum Regional Training & Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/10-106
Record Dates: First submitted 2020-05-22; First posted 2020-06-04 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2020-07

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Extracorporeal shock wave therapy; Carpal Tunnel Syndrome; physical therapy
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Splints; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: This study aims to compare the efficacy of RESWT to the recommended conventional PT modalities, including therapeutic US, in the treatment of CTS with regards to nociceptive and neuropathic pain, functionality and nerve conduction study outcomes.
Who Masked: Outcomes Assessor
Masking Description: All pre and post study evaluations will be performed by a single physical medicine and rehabilitation specialist blind to the patients' treatment groups. Patients will be randomised into the groups by a second physical medicine and rehabilitation specialist. PT wil be conducted by a single experienced physiotherapist. All data analysis will be conducted by a PMR specialist blind to the treatment provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group-1 splint and home exercise (Active Comparator): Patients in group 1 will be treated with splinting of the affected hand at night and a home exercise program. A wrist orthosis which held the wrist in the neutral position will be used for splinting at night time for a minimum of eight hours. Each patient will be given a home exercise program of wrist range of motion, wrist stretch, wrist isometric strengthening and median nerve glide exercises to be performed daily for the duration of the study
  Interventions: Device: splint and home exercise
- group 2 RESWT (Active Comparator): Patients in group 2 will be treated with splinting of the affected wrist at night, a home exercise program similar to that of group one and a total of 3 sessions of RESWT at a frequency of one session per week using the Masterpuls ® mp200 radial shock wave therapy system (Elite-Storz Medical AG, Kreuzlingen, Switzerland). RESWT at a pressure of 4 bars, a frequency of 5Hz and 2000 hits in total will be applied 2cm proximal to the median nerve, with the probe directed towards the palm, diffusely over the pisiform.
  Interventions: Device: RESWT
- group 3 physical therapy (Active Comparator): Patients in group 3 will be treated with splinting of the affected wrist at night, a home exercise program similar to that of group one and two and 20 minutes of liquid paraffin treatment of the hand, 1.5watt/cm2 therapeutic ultrasound applied to the volar surface of the wrist for 5 minutes and 20 minutes of transcutaneous electrical nerve stimulation (TENS) on five consecutive days of the week for a total of fifteen sessions over 3 weeks.
  Interventions: Device: physical therapy

INTERVENTIONS:
Device: splint and home exercise — Each patient will be given a home exercise program of wrist range of motion, wrist stretch, wrist isometric strengthening and median nerve glide exercises to be performed daily for the duration of the study
  Arms: group-1 splint and home exercise
Device: RESWT — RESWT at a pressure of 4 bars, a frequency of 5Hz and 2000 hits in total will be applied 2cm proximal to the median nerve, with the probe directed towards the palm, diffusely over the pisiform.
  Other Names: splint and home exercise
  Arms: group 2 RESWT
Device: physical therapy — 20 minutes of liquid paraffin treatment of the hand, 1.5watt/cm2 therapeutic ultrasound applied to the volar surface of the wrist for 5 minutes and 20 minutes of transcutaneous electrical nerve stimulation (TENS) on five consecutive days of the week for a total of fifteen sessions over 3 weeks
  Other Names: splint and home exercise
  Arms: group 3 physical therapy

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common of all entrapment syndromes with a prevalence of 1-5%. Electrodiagnostic testing is used to make a definite diagnosis. The mainstay of the pathophysiology of CTS includes mechanical damage to the median nerve due to build up of pressure in the carpal tunnel and nerve ischaemia. Physical therapy (PT) in particular is the conventional non-surgical treatment of choice in the management of mild to moderate CTS, resulting in pain reduction and improved function.

Extracorporeal shock wave therapy (ESWT) is a non invasive treatment method in which high frequency sound waves are applied to the body. The mechanism of action of ESWT in the treatment of CTS remains largely unknown.

Eventhough there are many therapeutic options in the treatment of mild to moderate CTS, there is no consensus on the most effective treatment (4). ESWT has become a desirable treatment option in recent years. However, due to small patients numbers in trials to date and a lack of placebo controlled studies, the efficacy of this treatment option is still under debate. This study aims to compare the efficacy of RESWT to the recommended conventional PT modalities, including therapeutic US, in the treatment of CTS with regards to nociceptive and neuropathic pain, functionality and nerve conduction study outcomes.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is the most common of all entrapment syndromes with a prevalence of 1-5%. CTS describes the compression of the median nerve as it travels through the carpal tunnel of the wrist, largely resulting in sensory symptoms of paraesthesia and pain in the areas of the hand innervated by the nerve. CTS can also lead to muscle atrophy, loss of motor function and disability of the hand. Electrodiagnostic testing is used to make a definite diagnosis. The mainstay of the pathophysiology of CTS includes mechanical damage to the median nerve due to build up of pressure in the carpal tunnel and nerve ischaemia. Chronic compression of the median nerve also results in neuronal depolarisation and the release of neuropeptides such as substance P and calcitonin-gene-related peptide. These neuropeptides stimulate the release of endothelial nitric oxide thus triggering vasodilatation and neurogenic inflammation .

Management of CTS depends on disease severity. Physical therapy (PT) in particular is the conventional non-surgical treatment of choice in the management of mild to moderate CTS, resulting in pain reduction and improved function. Recommended PT modalities include laser, ultrasound and liquid paraffin therapy. US therapy in particular has given satisfactory results in the treatment of mild to moderate CTS. The biophysical effects of US have been shown to trigger nerve regeneration and healing.

Extracorporeal shock wave therapy (ESWT) is a non invasive treatment method in which high frequency sound waves are applied to the body . ESWT can be divided into radial (RESWT) and focused (FESWT) based on the design of the reflector and resultant pressure and energy applied. Animal studies have shown that ESWT, and especially RESWT can be successfully used in the treatment of peripheral nerve lesions, improving nerve regeneration and functional activity . Human studies on its uses in the treatment of peripheral neuropathies such as interdigital neuroma, distally symmetric polyneuropathy and CTS have also given promising results . The mechanism of action of ESWT in the treatment of CTS remains largely unknown. However, it is believed that the antiinflammatory, angio- and neuro-genic, effects of ESWT encourages tissue regeneration in CTS thus reducing the patient's symptoms and promoting an improvement in function. Moreover, RESWT rather than FESWT maybe the better therapeutic option in CTS as it can be applied to a wider area, incorporating both the median nerve and surrounding tissues.

Eventhough there are many therapeutic options in the treatment of mild to moderate CTS, there is no consensus on the most effective treatment. ESWT has become a desirable treatment option in recent years. However, due to small patients numbers in trials to date and a lack of placebo controlled studies, the efficacy of this treatment option is still under debate. This study aims to compare the efficacy of RESWT to the recommended conventional PT modalities, including therapeutic US, in the treatment of CTS with regards to nociceptive and neuropathic pain, functionality and nerve conduction study outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients have symptoms of CTS for more than three months with physical examination and electrophysiological findings consistent with mild to moderate CTS

Exclusion Criteria:

1. Presence of other sensory or motor neuropathies
2. History of surgery, trauma or fracture of the index hand and wrist
3. History of corticosteroid injection or PT of the index wrist within the past three months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
The Boston carpal tunnel questionnaire (BCTQ) | Change from Baseline BCTQ at 3 weeks post-treatment
  This questionnaire determines symptom severity (BCTQs) and functional outcome (BCTQf) specific to CTS using a scale for each. BCTQs is determined using 11 questions each with 5 answers to choose from scored from 1 to 5 giving a BCTQs total out of 55. The higher the score the greater the symptom severity. BCTQf questions the difficulty of 8 functional activities scored from 1 to 5 giving a BCTQf total out of 40. The higher the score the worse the functional capacity

SECONDARY OUTCOMES:
Visual analogue scale (VAS) | Change from Baseline VAS at 3 weeks post-treatment
  The VAS provides a subjective, visual linear pain score from 0-10cm scored by the patient where 0cm is no pain (0cm is no pain and 10cm the worst pain imaginable)
Leeds Assesment of Neuropathic Symptoms and Signs (LANSS) | Change from Baseline LANSS at 3 weeks post-treatment
  LANSS is a bedside test used to differentiate between nociceptive and neuropathic pain. The first part of the LANSS consists of five questions on neuropathic pain (maximum score of 16). The second part is a physical examination performed by the physician to elicit neuropathic pain. A final test score of 12 and above signifies neuropathic pain, a score below 12 signifies nociceptive pain with a sensitivity of 83% and a specificity of 87%

CONTACTS AND LOCATIONS:
Overall Officials: Gonca Saglam, MD, Principal Investigator — Erzurum Regional Traning and
Locations (2):
- Turkey (Türkiye) (2):
  - Baskent University, Ankara
  - Erzurum Regional Training & Research Hospital, Erzurum

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after identification (text,tables,figures) will be made available
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Individual participant data that underlie the results reported in this article, after identification (text,tables,figures) will be made available
Access Criteria: The data will be shared with researchers providing a methodologically sound proposal. Proposals should be directed to goncasaglam@hotmail.com. To gain access , data requestors will need to sign a data access agreement. Data will be accessible for a period of one year.

REFERENCES:
- [Background] Kim JC, Jung SH, Lee SU, Lee SY. Effect of extracorporeal shockwave therapy on carpal tunnel syndrome: A systematic review and meta-analysis of randomized controlled trials. Medicine (Baltimore). 2019 Aug;98(33):e16870. doi: 10.1097/MD.0000000000016870. PMID 31415424
- [Background] Vahdatpour B, Kiyani A, Dehghan F. Effect of extracorporeal shock wave therapy on the treatment of patients with carpal tunnel syndrome. Adv Biomed Res. 2016 Jul 29;5:120. doi: 10.4103/2277-9175.186983. eCollection 2016. PMID 27563630
- [Background] Paoloni M, Tavernese E, Cacchio A, D'orazi V, Ioppolo F, Fini M, Santilli V, Mangone M. Extracorporeal shock wave therapy and ultrasound therapy improve pain and function in patients with carpal tunnel syndrome. A randomized controlled trial. Eur J Phys Rehabil Med. 2015 Oct;51(5):521-8. Epub 2015 Feb 20. PMID 25697763